CLINICAL TRIAL: NCT05971680
Title: the Effect of Vitamin B 1 on Menstrual Pattern After Insertion of the IUD.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vitamin B 1 IUD
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Intra-uterine Device Complication
Keywords: Intra-uterine Device; Vitamin B 1
MeSH Terms: interventions — Thiamine; Intrauterine Devices

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B 1 (Experimental): VITAMIN B1 (High Potency) 500mg
  Interventions: Drug: VITAMIN B1 500mg; Device: intra-uterine contraceptive device
- control (Other): patient not subjected to treatment . only follow up
  Interventions: Device: intra-uterine contraceptive device

INTERVENTIONS:
Drug: VITAMIN B1 500mg — VITAMIN B1 (High Potency) 500mg tab every day for 3 months
  Other Names: VITAMIN B1 500mg @Biovea
  Arms: Vitamin B 1
Device: intra-uterine contraceptive device — intra-uterine contraceptive device
  Other Names: silverline IUD

SUMMARY:
investigate the effect of vitamin B 1 on menstrual bleeding and spotting after insertion of the IUD.

DETAILED DESCRIPTION:
This study will be randomized controlled trial will be performed at the Obstetric and Gynecological Department at Beni-Suef University Hospital, Faculty of Medicine Target Population: All females with first time use of IUD inserted at the Obstetrics and Gynecology department through 3 months from the start of July 2023 till the end of November 2023.

Participants will be assigned in a 1:1 ratio to the use of vitamin B 1 or placebo, in accordance with a random table produced by an Excel program, with A being assigned to the intervention group and B to the control group. All women will sign a written informed consent prior to data collection.

Each woman within the intervention group will receive a packet containing 30 pills (vitamin B 1 or placebo), each month for three months.

ELIGIBILITY:
Inclusion Criteria:

* Females with first time use of the IUD
* a history of normal menstrual bleeding with duration of 3 to 7 days without spotting, a menstrual cycle lasting 23 to 35 days,
* use of 10 to 14 sanitary pads per cycle before IUD insertion
* gravidity ranging between 1 and 4.

Exclusion Criteria:

* Patients with cardiac, hepatic or renal diseases.
* Patients with bleeding disorders.
* Patients with systemic diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
the duration of menstrual bleeding. | 3 cycles ( 3 months / one month for each cycle)
  days of menstruation

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided